CLINICAL TRIAL: NCT04913220
Title: A Phase 1/2 Non-randomized, Open-label, Multi-cohort, Multi-center Study Assessing the Clinical Benefit of SAR444245 (THOR- 707) Combined With Cemiplimab for the Treatment of Participants With Advanced Unresectable or Metastatic Skin Cancers
Brief Title: A Study of SAR444245 Combined With Cemiplimab for the Treatment of Participants With Various Advanced Skin Cancers (Pegathor Skin 201)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early discontinuation based on strategic sponsor decision not driven by any safety concerns
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT16845; U1111-1254-0189 (Registry Identifier: ICTRP); 2020-005332-30 (EudraCT Number)
Record Dates: First submitted 2021-05-28; First posted 2021-06-04 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Malignant Melanoma; Squamous Cell Carcinoma of Skin
MeSH Terms: conditions — Melanoma | interventions — cemiplimab; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Melanoma (Experimental): SAR444245 and cemiplimab administered every 3 weeks on Day 1 of each cycle (21 days per cycle) for up to 35 cycles.
  Interventions: Drug: THOR-707; Drug: Cemiplimab
- Cohort B: cutaneous squamous cell carcinoma (CSCC) (Experimental): SAR444245 and cemiplimab administered every 3 weeks on Day 1 of each cycle (21 days per cycle) for up to 35 cycles.
  Interventions: Drug: THOR-707; Drug: Cemiplimab

INTERVENTIONS:
Drug: THOR-707 — Solution for infusion: intravenous infusion
Drug: Cemiplimab — Solution for infusion: intravenous infusion
  Other Names: Libtayo® or generic

SUMMARY:
Primary Objective:

-To determine the antitumor activity of SAR444245 in combination with cemiplimab.

Secondary Objectives:

* To determine the recommended phase 2 dose and to assess the safety profile of SAR444245 when combined with cemiplimab
* To assess other indicators of antitumor activity
* To assess the concentrations of SAR444245 when given in combination with cemiplimab
* To assess the immunogenicity of SAR444245
* To assess active concentrations of cemiplimab when given in combination with SAR444245

DETAILED DESCRIPTION:
The duration of the study for an individual patient will start from the signature of the main informed consent and include a screening period of up to 28 days, a treatment period [max 35 cycles or until PD], an end-of-treatment visit 30 days + 7 days following the last administration of study drug (or until the patient receives another anticancer therapy, whichever is earlier), and a follow-up visit 3 months after treatment discontinuation and every 3 months following, until disease progression, or initiation of another antitumor treatment, or final cohort cut-off, whichever is earlier

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age (or country's legal age of majority if >18 years), at the time of signing the informed consent.
* Participants with:
* Cohort A: Histologically confirmed unresectable locally advanced or metastatic melanoma that are not amenable to local therapy
* Cohort B: Histologically confirmed metastatic CSCC or locally advanced
* CSCC that are not candidates for curative surgery or radiation. Special considerations for the following categories:

Participants with tumors arising on the cutaneous hair (non-glabrous) bearing lip with extension onto dry red lip (vermillion) may be eligible after communication with and approval from the Sponsor

Participants with the primary site is nose are only eligible if the primary site was skin, not nasal mucosa with outward extension to skin (the Investigator confirmed)

Participants with mixed histology in which the predominant histology is invasive CSCC may be eligible after communication with and approval from the Sponsor

* Participants in both cohorts must have at least one measurable lesion
* Provision of tumor tissue:

For participants in the dose escalation:

16 µg/kg: at screening, biopsy is optional but highly recommended; and on-treatment not required

24 µg/kg: at screening, biopsy is mandatory and on-treatment, optional but highly recommended

* For the other participants : Mandatory baseline biopsy for the participants to enroll in cohort A with skin metastasis and in cohort B. Mandatory on-treatment biopsy for participants in Cohort A with skin metastasis and participants in Cohort B.
* Females are eligible to participate if they are not pregnant or breastfeeding, not a woman of childbearing potential (WOCBP) or are a WOCBP that agrees: to use approved contraception method and submit to regular pregnancy testing prior to treatment and for at least 180 days after discontinuing study treatment and to refrain from donating or cryopreserving eggs for 180 days after discontinuing study treatment.
* Males are eligible to participate if they agree to refrain from donating or cryopreserving sperm, and either abstain from heterosexual intercourse OR use approved contraception during study treatment and for at least 210 days after discontinuing study treatment.
* Capable of giving signed informed consent

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:
* Eastern Cooperative Oncology Group (ECOG) performance status of ≥2
* Poor organ function
* Participants with baseline SpO2 ≤92%
* Active brain metastases or leptomeningeal disease.
* History of allogenic tissue/solid organ transplant.
* Last administration of prior antitumor therapy or any investigational treatment within 28 days or less than 5 times the half-life, whichever is shorter; major surgery or local intervention within 28 days.
* History of lung disease
* Comorbidity requiring corticosteroid therapy
* Antibiotic use (excluding topical antibiotics) ≤14 days prior to first dose of IMP
* Severe or unstable cardiac condition within 6 months prior to starting study treatment
* Active, known, or suspected autoimmune disease that has required systemic treatment in the past 2 years
* Known second malignancy either progressing or requiring active treatment within the last 3 years

For both cohorts:

* Prior immune checkpoint inhibitors except in the context of adjuvant or neoadjuvant; Participants who were on control arm of a study with an investigational anti-PD-1/PD-L1 are eligible.
* Received adjuvant or neoadjuvant therapy during the 6 months prior to development of metastatic disease.
* For Cohort A: any prior systemic treatment for advanced/metastatic disease
* For Cohort B: >2 prior lines of any systemic treatment for advanced/metastatic disease
* Inability to undergo any contrast-enhanced radiologic response assessment
* Receipt of a live-virus vaccination within 28 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2025-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- Beverly Hills Cancer Center & Optima Diagnostic Imaging Site Number : 8400007, Beverly Hills, California, United States
- Investigational Site Number : 0360001, Macquarie University, New South Wales, Australia
- Chile (6):
  - Investigational Site Number : 1520005, Santaigo, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Antofagasta
  - Investigational Site Number : 1520003, Temuco
- France (5):
  - Investigational Site Number : 2500003, Bobigny
  - Investigational Site Number : 2500002, Dijon
  - Investigational Site Number : 2500005, Lille
  - Investigational Site Number : 2500001, Nantes
  - Investigational Site Number : 2500006, Pierre-Bénite
- Germany (5):
  - Investigational Site Number : 2760004, Berlin
  - Investigational Site Number : 2760001, Hamburg
  - Investigational Site Number : 2760003, Mannheim
  - Investigational Site Number : 2760006, Minden
  - Investigational Site Number : 2760005, München
- Italy (2):
  - Investigational Site Number : 3800001, Napoli
  - Investigational Site Number : 3800004, Perugia
- Spain (4):
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240004, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240002, Santander, Cantabria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT16845 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25199&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 21 centers (corresponds to number of sites which screened at least one participant) in 7 countries. Out of 61 participants who were screened from 15 July 2021 to 25 October 2022, 46 participants were enrolled in the study.
Pre-assignment Details: The study was terminated based on strategic sponsor decision not driven by any safety concerns.
  Note: Reason for not completed = Reason for permanent full intervention discontinuation.
Groups:
- Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab: Participants who were immune checkpoint inhibitor (ICI)- naïve and previously untreated locally advanced, unresectable or metastatic melanoma were included in this cohort. Participants received pegenzileukin 16 microgram per kilogram (mcg/kg) along with cemiplimab 350 milligram (mg) via intravenous (IV) infusion over 30 minutes every 3 weeks (q3w) on Day 1 of each cycle (each cycle is 21 days) (as first-line [1L] therapy), until disease progression (PD), unacceptable adverse event (AE) or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab: Participants who were ICI- naïve and previously untreated locally advanced, unresectable or metastatic melanoma were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with cemiplimab 350 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 1L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab: Participants with ICI-naïve, metastatic or locally advanced cutaneous squamous cell carcinoma (CSCC) who were not candidates for curative surgery or curative radiation and who received no more than 2 prior lines of systemic therapy were included in this cohort. Participants received pegenzileukin 16 mcg/kg along with cemiplimab 350 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as first to third line [1-3L] therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab: Participants with ICI-naïve, metastatic or locally advanced CSCC who were not candidates for curative surgery or curative radiation and who received no more than 2 prior lines of systemic therapy were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with cemiplimab 350 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 1-3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
Period: Overall Study
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Started | 20 | 7 | 16 | 3
Completed | 4 | 2 | 4 | 0
Not Completed | 16 | 5 | 12 | 3
Not completed — Not Related to Coronavirus Disease 2019 (COVID-19) | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 0
Not completed — Poor Compliance to Protocol | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 8 | 4 | 3 | 2
Not completed — Adverse event: Not related to COVID-19 | 7 | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Population: The exposed population consisted of all participants who had given their informed consent and received at least one dose of study treatment.
Groups:
- Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab: Participants who were ICI- naïve and previously untreated locally advanced, unresectable or metastatic melanoma were included in this cohort. Participants received pegenzileukin 16 mcg/kg along with cemiplimab 350 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 1L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab: Participants with ICI-naïve, metastatic or locally advanced CSCC who were not candidates for curative surgery or curative radiation and who received no more than 2 prior lines of systemic therapy were included in this cohort. Participants received pegenzileukin 16 mcg/kg along with cemiplimab 350 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 1-3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Total: Total of all reporting groups
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Total
Number analyzed (Participants) | 20 | 7 | 16 | 3 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (11.7) | 56.1 (12.9) | 69.8 (14.3) | 74.0 (21.0) | 64.2 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 5 | 0 | 15
  Male | 13 | 4 | 11 | 3 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 20 | 6 | 13 | 2 | 41
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 3 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: All Cohorts: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of participants who had best overall response (BOR) as confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 or modified world health organization (WHO) response criteria. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 millimeter (mm) (<1 centimeter [cm]). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to approximately 25 months (Cohorts A and B)
Population: The efficacy population consisted of all participants from the exposed population with at least one evaluable post-baseline tumor assessment or who permanently discontinued study treatment.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 20 | 7 | 16 | 3
Percentage of participants | 40.0 [21.7 to 60.6] | 57.1 [22.5 to 87.1] | 56.3 [33.3 to 77.3] | 0 [0.0 to 63.2]

2. Secondary Outcome: All Cohorts: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was any AE that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were defined as AEs that developed, worsened (according to the investigator's opinion) or became serious during the TE period.
Time Frame: From first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment; approximately 27 months (Cohorts A and B)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 20 | 7 | 16 | 3
Participants
  TEAEs | 20 | 7 | 16 | 3
  TESAEs | 11 | 4 | 8 | 1

3. Secondary Outcome: All Cohorts: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Selected events that occurred during the DLT observation period were considered as DLT unless due to PD or to a cause obviously unrelated to pegenzileukin. Selected events included: any grade 4 neutropenia irrespective of duration; any febrile neutropenia; grade 3 thrombocytopenia associated with transfusion in addition to bleeding and any grade 4 thrombocytopenia; grade 3 or above: alanine aminotransferase or aspartate aminotransferase, vascular leak syndrome, hypotension, cytokine release syndrome, and AE that did not resolve to grade <=2 within 7 days of starting accepted standard of care medical management; and grade 4 laboratory abnormalities.
Time Frame: From Day 1 to Day 21 of Cycle 1 (each cycle is 21 days: Cohorts A and B)
Population: The DLT-evaluable population consisted of all exposed participants in the dose escalation who had been treated and observed for at least 21 days. Any participants who had experienced a DLT during DLT observation period were also DLT-evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 5 | 7 | 4 | 3
Participants | 1 | 1 | 1 | 1

4. Secondary Outcome: All Cohorts: Complete Response (CR) Rate
Description: The CR rate was defined as the percentage of participants who had a confirmed CR as per RECIST v 1.1 or modified WHO response criteria. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm).
Time Frame: From first dose of study treatment administration (Day 1) up to maximum exposure of study treatment, approximately 26 months (Cohorts A and B)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 20 | 7 | 16 | 3
Percentage of participants | 5.0 [0.3 to 21.6] | 14.3 [0.7 to 52.1] | 0 [0.0 to 17.1] | 0 [0.0 to 63.2]

5. Secondary Outcome: All Cohorts: Time to Complete Response
Description: The time to CR was defined as the time from the first administration of study treatment to the first tumor assessment at which the overall response was recorded as CR that was subsequently confirmed as per RECIST v 1.1 or modified WHO response criteria. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm).
Time Frame: as for outcome 4
Population: The efficacy population consisted of all participants from the exposed population with at least one evaluable post-baseline tumor assessment or who permanently discontinued study treatment. Only participants with confirmed CR were analyzed.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 1 | 1 | 0 | 0
Months | 4.0 [4 to 4] | 4.0 [4 to 4] |  |

6. Secondary Outcome: All Cohorts: Time to Response (TTR)
Description: The TTR was defined as the time from the first study treatment administration to the first tumor assessment at which the overall response was recorded as PR or CR that was subsequently confirmed as per RECIST v 1.1 or modified WHO response criteria. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 4
Population: The efficacy population consisted of all participants from the exposed population with at least one evaluable post-baseline tumor assessment or who permanently discontinued study treatment. Only participants with confirmed CR or PR were analyzed.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 8 | 4 | 9 | 0
Months | 2.1 [2 to 6] | 2.1 [2 to 4] | 2.8 [2 to 4] |

7. Secondary Outcome: All Cohorts: Duration of Response (DOR)
Description: The DOR was defined as the time from the first tumor assessment at which the overall response was recorded as CR or PR that was subsequently confirmed until documented PD before the initiation of any subsequent anti-cancer therapy or death due to any cause, whichever occurred first, as per RECIST v 1.1 or modified WHO response criteria. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study), in addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm (0.5 cm).
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 8 | 4 | 9 | 0
Months | NA [8.5 to NA] — NA indicates that the median and upper limit of 90% confidence interval (CI) was not estimable due to insufficient number of participants with events. | NA [4.2 to NA] — NA indicates that the median and upper limit of 90% CI was not estimable due to insufficient number of participants with events. | NA [4.1 to NA] — NA indicates that the median and upper limit of 90% CI was not estimable due to insufficient number of participants with events. |

8. Secondary Outcome: All Cohorts: Clinical Benefit Rate (CBR)
Description: The CBR was defined as the percentage of participants with clinical benefit: confirmed CR or PR as BOR, or stable disease (SD) lasting at least 6 months, as per RECIST v 1.1 or modified WHO response criteria. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. BOR was defined as the best response observed from the start of the study treatment until PD, death, cut-off date or initiation of post-treatment anti-cancer therapy, whichever occurred first. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 20 | 7 | 16 | 3
Percentage of participants | 40.0 [21.7 to 60.6] | 57.1 [22.5 to 87.1] | 56.3 [33.3 to 77.3] | 0 [0.0 to 63.2]

9. Secondary Outcome: All Cohorts: Progression Free Survival (PFS)
Description: The PFS was defined as the time from the date of first study treatment administration to the date of the first documentation of objective PD, or death due to any cause, whichever occurred first, as per RECIST v 1.1 or modified WHO response criteria. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study), in addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm (0.5 cm).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 20 | 7 | 16 | 3
Months | 6.2 [2.1 to NA] — NA indicates that the upper limit of 90% CI was not estimable due to insufficient number of participants with events. | 6.2 [2.0 to NA] — NA indicates that the upper limit of 90% CI was not estimable due to insufficient number of participants with events. | NA [4.1 to NA] — NA indicates that the median and upper limit of 90% CI were not estimable due to insufficient number of participants with events. | 4.2 [4.1 to NA] — NA indicates that the upper limit of 90% CI was not estimable due to insufficient number of participants with events.

10. Secondary Outcome: All Cohorts: Plasma Concentrations of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of plasma concentrations of pegenzileukin.
Time Frame: Cycle 1 Days 2 and 3 (each cycle is 21 days)
Population: The pharmacokinetic (PK) population consisted of all participants from exposed population with at least one PK concentration available after the first dose of study treatment. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 20 | 7 | 14 | 2
Nanograms per milliliter (ng/mL)
  Cycle 1 Day 2 | 114.6 (48.7) | 209.4 (58.3) | 105.2 (33.8) | 137.0 (15.6)
  Cycle 1 Day 3: number analyzed (Participants) | 5 | 6 | 4 | 2
  Cycle 1 Day 3 | 26.1 (13.8) | 74.4 (22.0) | 31.1 (11.3) | 61.4 (18.4)

11. Secondary Outcome: All Cohorts: Number of Participants With Anti-Drug Antibodies (ADAs) Against Pegenzileukin
Description: Blood samples were collected at specified timepoints to assess the presence of ADAs against pegenzileukin. Treatment-emergent ADA was defined as at least one treatment-induced or treatment-boosted ADA. Treatment-induced ADA was defined as ADA that developed during the TE period and without pre-existing ADA (including participants without pre-treatment samples). Treatment-boosted ADA was defined as pre-existing ADA that was boosted during the TE period to a significant higher titer than the baseline. Number of participants with treatment-emergent ADA is presented.
Time Frame: as for outcome 2
Population: The ADA population consisted of all participants from the exposed population with at least one ADA result (positive, negative or inconclusive) after the first dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 20 | 7 | 12 | 3
Participants | 0 | 1 | 1 | 0

12. Secondary Outcome: All Cohorts: Concentration Observed Just Before Study Treatment Administration During Repeated Dosing (Ctrough) of Cemiplimab
Description: Blood samples were collected at specified timepoints for the assessment of Ctrough of cemiplimab. The PK population consisted of all participants from exposed population with at least one PK concentration available after the first dose of study treatment. Only participants with data collected at specified timepoints are reported.
Time Frame: Cycles 1, 2, 4, 7, 10, and 15 (each cycle is 21 days)
Population: Eventually, the participants discontinued as they progressed in the study. Hence, fewer participants at each cycle and no participants returned i.e. no sample was collected for Cycle 10 for Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab and Cycle 15 for Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab and Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 19 | 7 | 14 | 3
ng/mL
  Cycle 1 | 47.6 (207.6) | 901.4 (1965.0) | 0.0 (0.0) | 0.0 (0.0)
  Cycle 2: number analyzed (Participants) | 15 | 7 | 12 | 2
  Cycle 2 | 14368.0 (4519.9) | 20685.7 (8170.6) | 24215.8 (30639.3) | 24200.0 (12445.1)
  Cycle 4: number analyzed (Participants) | 10 | 6 | 8 | 1
  Cycle 4 | 37028.0 (26202.1) | 43383.3 (19397.5) | 37112.5 (19946.6) | 8310.0 (NA) — NA indicates that the standard deviation (SD) was not estimable for 1 participant.
  Cycle 7: number analyzed (Participants) | 3 | 5 | 4 | 1
  Cycle 7 | 47333.3 (24339.5) | 59500.0 (30389.6) | 50825.0 (12601.7) | 23500.0 (NA) — NA indicates that the SD was not estimable for 1 participant.
  Cycle 10: number analyzed (Participants) | 2 | 3 | 4 | 0
  Cycle 10 | 40300.0 (1697.1) | 55933.3 (17201.6) | 67050.0 (22657.2) |
  Cycle 15: number analyzed (Participants) | 1 | 0 | 4 | 0
  Cycle 15 | 45900.0 (NA) — NA indicates that the SD was not estimable for 1 participant. |  | 58075.0 (15320.0) |

13. Secondary Outcome: All Cohorts: Concentration at End of Infusion (Ceoi) of Cemiplimab
Description: Blood samples were collected at specified timepoints for the assessment of Ceoi of cemiplimab. The PK population consisted of all participants from exposed population with at least one PK concentration available after the first dose of study treatment. Only participants with data collected at specified timepoints are reported.
Time Frame: Cycles 1, 2, 4, 7, 10, and 15 (each cycle is 21 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
Number analyzed (Participants) | 19 | 7 | 14 | 2
ng/mL
  Cycle 1 | 73494.7 (34263.7) | 90500.0 (32177.0) | 83857.1 (29231.3) | 92550.0 (9970.2)
  Cycle 2: number analyzed (Participants) | 15 | 7 | 12 | 2
  Cycle 2 | 98026.7 (15015.6) | 56142.9 (31838.5) | 108025.0 (30238.6) | 143500.0 (707.1)
  Cycle 4: number analyzed (Participants) | 10 | 6 | 8 | 1
  Cycle 4 | 107670.0 (45761.5) | 93683.3 (34262.9) | 130487.5 (46562.0) | 113000.0 (NA) — NA indicates that the SD was not estimable for 1 participant.
  Cycle 7: number analyzed (Participants) | 3 | 5 | 4 | 1
  Cycle 7 | 108833.3 (20336.7) | 125260.0 (38195.4) | 149000.0 (28248.9) | 137000.0 (NA) — NA indicates that the SD was not estimable for 1 participant.
  Cycle 10: number analyzed (Participants) | 2 | 3 | 4 | 0
  Cycle 10 | 121500.0 (6364.0) | 91166.7 (29458.8) | 171000.0 (48996.6) |
  Cycle 15: number analyzed (Participants) | 1 | 0 | 4 | 0
  Cycle 15 | 129000.0 (NA) — NA indicates that the SD was not estimable for 1 participant. |  | 159250.0 (17231.3) |

ADVERSE EVENTS:
Time Frame: Adverse events data was collected from first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment; approximately 27 months (Cohorts A and B). All-cause mortality (death) was assessed from first dose of study treatment (Day 1) up to end of follow-up for each participant, approximately 43 months.
Description: Analysis was performed on the exposed population.
Arm/Group | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab
All-Cause Mortality (participants affected / at risk) | 5/20 | 2/7 | 2/16 | 0/3
Serious Adverse Events (participants affected / at risk) | 11/20 | 4/7 | 8/16 | 1/3
Other Adverse Events (participants affected / at risk) | 19/20 | 7/7 | 16/16 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab (N=20) | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab (N=7) | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab (N=16) | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab (N=3)
Abdominal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Immune-Mediated Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningoradiculitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myasthenic Syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-Mediated Myocarditis (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric Antral Vascular Ectasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-Mediated Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-Mediated Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-Mediated Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prerenal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (11) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab (N=20) | Cohort A:1L Melanoma ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab (N=7) | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 16 mcg/kg + Cemiplimab (N=16) | Cohort B: 1-3L CSCC ICI-naïve: Pegenzileukin 24 mcg/kg + Cemiplimab (N=3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suspected Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 3 (6) | 1 (2) | 2 (4) | 1 (1)
Glucocorticoid Deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperadrenocorticism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Immune-Mediated Adrenal Insufficiency (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Immune-Mediated Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-Mediated Hypothyroidism (Endocrine disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 3 (6) | 1 (1) | 3 (4) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (9) | 2 (4) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (6) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Immune-Mediated Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tension Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Macular Neuroretinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 0 (0) | 3 (4) | 1 (2)
Systolic Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Immune-Mediated Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 2 (4) | 3 (4) | 1 (2)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (3) | 4 (5) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Immune-Mediated Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-Mediated Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8) | 1 (1) | 4 (4) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 2 (2) | 0 (0)
Rash Macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Immune-Mediated Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (12) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 4 (5) | 4 (9) | 2 (5) | 1 (1)
Chills (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Facial Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (4) | 0 (0) | 6 (7) | 1 (1)
Influenza Like Illness (General disorders) | 0 (0) | 3 (16) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Amylase Increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
Blood Albumin Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood Calcium Decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Blood Chloride Increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Magnesium Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Phosphorus Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Triglycerides Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Urea Increased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
C-Reactive Protein Increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cortisol Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase Increased (Investigations) | 1 (1) | 1 (7) | 2 (3) | 0 (0)
Procalcitonin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein Total Decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Prothrombin Time Prolonged (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 13 (53) | 5 (12) | 14 (86) | 2 (7)
Skin Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated based on strategic sponsor decision not driven by any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT04913220/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT04913220/SAP_001.pdf